UAN: 042-111-747-424 www.riphah.edu.pk 048567

## Research & Ethics Committee

RIPHAH INTERNATIONAL UNIVERSITY Educate triughten Empower

Riphah College of Rehabilitation and Allied Health Sciences Faculty of Rehabilitation and Allied Health Sciences Riphah International University, Lahore, Pakistan

Ref. No. REC/RCR & AHS/23/1103

Date: March 07, 2023

## TO WHOM IT MAY CONCERN

SUBJECT: INSTITUTIONAL APPROVAL OF THE RESEARCH STUDY

It is certified that Ms. Muzna Munir, Roll/Reg No.: 9841 is a bonafide student of Riphah College of Rehabilitation and Allied Health Sciences, Riphah International University, Lahore. She is enrolled in a doctorate degree program "Doctor of Philosophy in Rehabilitation Sciences". On behalf of Research and Ethics Committee (REC) it is to inform that the submitted research proposal entitled "Effects of supervised structured aerobic exercise training program on serum BDNF, androgens level, menstrual irregularity and quality of life in females with insulin resistant polycystic ovarian syndrome" has been reviewed and conforms to the REC guidelines. The Committee recommends that the proposal be commenced as planned.

Please note that this approval is valid for a period of two years only from the date of issuance and will require fresh approval if the study requires any change in the proposal or extension in the duration. It is advised to submit a revised protocol to REC for prior approval. It is emphasized that the study be conducted strictly in accordance with the submitted proposal.

Yours sincerely,

Research & Ethical Review Committee Righah College of Rehab. & Allied Health Sciences Righah International University Lahore

Muneeb-Khan, Ph.D.

Secretary

Research and Ethics Committee

Riphah College of Rehabilitation and Allied Health Sciences

Riphah International University, Lahore, Pakistan

Email: research.frahslhr@riphah.edu.pk